CLINICAL TRIAL: NCT04954911
Title: Prospective, Multi-centre, Observational Registry to Evaluate the Clinical Performance of the Globe® Mapping and Ablation System for the Treatment of Atrial Fibrillation
Brief Title: Clinical Performance of the Globe® Mapping and Ablation System for the Treatment of Atrial Fibrillation
Acronym: GLOBE-EU
Status: Completed | Type: Observational
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOC-138528
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Radiofrequency RF Ablation; Globe Mapping and Ablation System
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, multicentre, prospective, post-market product registry for participants with AF for whom ablation by the commercially available Globe Mapping and Ablation System was indicated before enrolment into the registry. The aim of the registry is to confirm the clinical performance and safety of the Globe Mapping and Ablation System in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Participants with a documented history of atrial fibrillation indicated for ablation using the Globe Mapping and Ablation System before enrolment into registry
3. Signed informed consent

Exclusion Criteria:

1. Contraindication for catheter ablation with the Globe System
2. Participant is currently participating in an investigational study that would interfere with registry endpoints according to the participating physician's discretion.
3. Physical or mental condition because of which, in the opinion of the physician, the participant is not able to give informed consent or comply with physician instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age 18 years or older
  2. Participants with a documented history of atrial fibrillation indicated for ablation using the Globe Mapping and Ablation System before enrolment into registry
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Freedom from AF at 12 months following ablation with the Globe System | Up to 1 year
Freedom from AF/AFL/AT at 12 months following ablation with the Globe System | Up to 1 year
Device- and procedure-related adverse events within 12 months following ablation with the Globe System | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Herz- und Diabeteszentrum NRW, Principal Investigator — Klinik für Elektrophysiologie/Rhythmologie Herz- und Diabeteszentrum NRW Universitätsklinik der Ruhr-Universität Bochum
Locations (2):
- Germany (2):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum Leipzig, Leipzig, Saxony